CLINICAL TRIAL: NCT06321770
Title: Oral Supplementation With Low Molecular Weight Collagen Peptides Improves Facial Wrinkles and Skin Hydration: Results From a Six-Week Randomized, Double-Blind, Placebo-Controlled Study
Brief Title: Oral Supplementation With Active Collagen Peptides and Skin Health Improvement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gala Servicios Clinicos S.L. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 075-2022
Record Dates: First submitted 2024-03-09; First posted 2024-03-20 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-03

CONDITIONS: Facial Wrinkles; Skin Hydration
Keywords: low molecular weight collagen peptides; aging; skin health; wrinkles; moisturization; elasticity; nutraceutical; randomized controlled trial

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind, Placebo-Controlled Study
Who Masked: Participant, Investigator
Masking Description: Randomized, Double-Blind, Placebo-Controlled Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bioactive collagen peptide (Experimental): The active treatment group included 40 women who received the bioactive collagen peptide-based food supplement orally
  Interventions: Dietary Supplement: Bioactive collagen peptides
- Placebo (Placebo Comparator): Oral suspension and sealed in sachets that were identical in appearance and odor.
  ingredients, which were also contained in the placebo, were 467 mg lemon flavour, 150 mg citric acid, 8.5 mg sucralose and 7.1 mg stevia (97%). The placebo did not contain any nutrients.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Bioactive collagen peptides — 2,5 g collagen peptides
  Arms: Bioactive collagen peptide
Dietary Supplement: Placebo — Placebo sachet daily
  Arms: Placebo

SUMMARY:
The present study aims to investigate the efficacy of daily supplementation with COLLinstant® LMW over a 6-week period in improving visible signs of aging. This in-cludes assessing its impact on skin wrinkle reduction, as well as its potential to en-hance skin elasticity and moisturization. COLLinstant® LMW was administered orally in a single-center, randomized, double-blind, placebo-controlled clinical trial. A sec-ondary objective involves comparing skin improvement, product satisfaction, and monitoring adverse events among middle-aged female volunteers.

DETAILED DESCRIPTION:
Study design and ethical aspects This was a 6-week, prospective, randomized, placebo-controlled, double-blind, monocentric study performed at GALA Laboratories in Don Benito-Villanueva (Badajoz, Spain).

Participants were individually randomized (1:1 ratio) to a strategy of receiving either COLLinstant® LMW (collagen group) or a placebo regimen and followed up for 6 weeks. Subjects were instructed to dose both product regimens as per the manufacturer's package instructions or, when appropriate, investigator guidance.

The investigation was performed according to the ethical guidelines detailed in the Declaration of Helsinki (amendment of the 64th General Assembly, Fortaleza, Brazil, October 2013) and with national regulations of Spain, and in full compliance with the applicable principles of good clinical practice (GCP) and International Council for Harmonisation (ICH) of Technical Requirements for Pharmaceuticals for Human Use. The trial protocol was approved (code 075-2022) by the Clinical Research Ethics Committee at the University Hospital of Cáceres (Caceres, Spain) and written informed consent was obtained from all subjects prior to any study procedures being ini-tiated.

Intervention/study products The test product is classified as a food supplement. The preparation under study was COLLinstant® LMW (Viscofan DE GmbH, Weinheim, Germany), an oral food supplement based on bovine bioactive hydrolyzed type I and III-collagen peptides.

Following ICH-GCP requirements and applicable local regulations, the inves-tigational product and placebo were presented as a powder for oral suspension and sealed in sachets that were identical in appearance and odor.

Each sachet of the active COLLinstant® LMW contained low molecular weight hydrolyzed 2.5 g collagen peptides. Other ingredients, which were also contained in the placebo, were 467 mg lemon flavour, 150 mg citric acid, 8.5 mg sucralose and 7.1 mg stevia (97%). The placebo did not contain any nutrients.

Study subjects We recruited a total of 80 women (aged 30-65 years) with phototypes I-IV, who were mentally and physically healthy, had a BMI 20.0-29.9 kg/m2 and displayed visible signs of natural and photoaging on their face (crow´s feet) rated from moderate to se-vere [21].

The Fitzpatrick scale is a numerical classification for human skin color (in a scale of I-VI), with the amount of melanin in the skin indicating the type of skin, its suscep-tibility to burns and its ability to tan.

During the screening phase, the participants satisfied all inclusion and exclusion criteria and agreed to avoid prolonged exposure to ultraviolet (UV) radiation for the duration of the study.

Subjects were excluded in case of pregnancy, lactation, acute or chronic skin dis-ease or dermatological disorder; use of natural health supplements for improving the skin within 1 month before the start of the study; low protein diet; planned or una-voidable exposure to UV radiation; tattoos on or near the test area; use of systemic cor-ticosteroids or applied topical alpha hydroxyl acids near the test site within 4 weeks of enrolment; use of topical medications near the test area within 6 weeks of enrolment; Botulinum toxin A (Botox) treatment or filler injection (collagen, hyaluronic acid, etc) near the test sites within 2 years of enrolment; subjects cognitively impaired and/or unable to give informed consent; or had any other condition which in the medical in-vestigator's opinion may adversely affect the individual's ability to complete the study or its measures or which may pose significant risk to the individual.

Study schedule and biometric evaluation All participants (test and placebo group) were instructed to consume the content of one sachet daily, in the morning, on an empty stomach for 6 weeks. It was required that the product was dissolved in at least 100 ml of water, juice or other liquid.

For all women participating in the study, biometric characteristics were assessed at baseline (T0), and after 6 weeks of treatment with the products (T6).

Measurement of skin wrinkling parameters (volume, area and depth) was evalu-ated at the crow's feet region and changes were analyzed and digitally photographed in all patients by VisioFace® 1000D (equipped with a high-resolution reflex camera).

Afterwards, subjects were acclimatized for at least 30 min in the air-conditioned measurement room at a temperature of 21 ± 1°C and a relative humidity of 50 ± 5 %.

Skin elasticity was measured at the crow's feet region, so a Cutometer® dual MPA 580 (Courage & Khazaka) was used to assess skin biomechanical properties. This non-invasive tool evaluated the skin elasticity by negative force that distorts the skin mechanically. The functional principle is based on suction of the skin using a probe with negative pressure (450 mbar), which causes the test area to be drawn into the ap-erture of the probe. A non-contact optical measuring system determined the penetra-tion depth of the skin. The parameters evaluated were R0, R2, R5, R7 y R9 and measurements were carried out in triplicate.

R0 represents the final distension of the first curve i.e., the passive behavior of the skin to the suction force and correlates to the skin firmness. This parameter is meas-ured from the highest point of amplitude at the end of the suction phase to the baseline reading (R0 = Uf).

The R2 parameter is related to the gross elasticity/ viscoelasticity, which is the skin's resistance to the mechanical suction force versus its ability to recover (R2 = Ua/Uf).

R5 refers to net elasticity and is represented by the ratio of the elastic portion of the suction stage to fast recovery throughout relaxation stage (R5 = Ur/Ue), meaning the higher the value, the more elastic the skin. R7 is related to biological elasticity. R7 is the immediate elastic recovery in the first 0.1 s compared with the amplitude (total deformation) after suction (R7 = Ur/Uf) and can be interpreted as another marker of elasticity, with aging causing its reduction; and R9, the residual deformation at the end of the measuring cycle, indicating the tiring effects or fatigue of skin after repeated suction (R9 = R3 - R0).

In addition, measurement of stratum corneum hydration was performed at each study visit by the electrical capacitance method using a Corneometer® CM 825 (Courage & Khazaka, Cologne, Germany). At least five determinations per measure-ment area at four different locations (middle forehead, both right and left cheek bone and the chin area) were performed, then the average was used for analysis.

Self-reported measures After 6 weeks of treatment, the volunteers filled out questionnaires, to subjectively assess their perception of different parameters such as efficacy, organoleptic properties and satisfaction since the last time they took the product. The Spanish version of the Treatment Satisfaction Questionnaire with Medication (TSQM), and a 3-point Likert scale with the following items: Dissatisfied, slightly satisfied and very satisfied, were used.

ELIGIBILITY:
Inclusion Criteria:

* Women (aged 30-65 years) with phototypes I-IV, who were mentally and physically healthy, had a BMI 20.0-29.9 kg/m2 and displayed visible signs of natural and photoaging on their face (crow´s feet) rated from moderate to severe

Exclusion Criteria:

* Pregnancy, lactation, acute or chronic skin disease or dermatological disorder; use of natural health supplements for improving the skin within 1 month before the start of the study; low protein diet; planned or unavoidable exposure to UV radiation; tattoos on or near the test area; use of systemic corticosteroids or applied topical alpha hydroxyl acids near the test site within 4 weeks of enrolment; use of topical medications near the test area within 6 weeks of enrolment; Botulinum toxin A (Botox) treatment or filler injection (collagen, hyaluronic acid, etc) near the test sites within 2 years of enrolment; subjects cognitively impaired and/or unable to give informed consent; or had any other condition which in the medical investigator's opinion may adversely affect the individual's ability to complete the study or its measures or which may pose significant risk to the individual.

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women aged 30 to 60 years
Enrollment: 80 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-04-16 (Actual); Study Completion 2024-06-03 (Actual)

PRIMARY OUTCOMES:
Skin wrinkling volume (px^3) | 6 weeks
  Measurement of skin wrinkling volume (px^3) was evaluated at the crow's feet region and changes were analyzed and digitally photographed in all patients by VisioFace® 1000D (equipped with a high-resolution reflex camera)
Skin wrinkling area (px^2) | 6 weeks
  Measurement of skin wrinkling area (px^2) was evaluated at the crow's feet region and changes were analyzed and digitally photographed in all patients by VisioFace® 1000D (equipped with a high-resolution reflex camera)
Skin wrinkling depth (px) | 6 weeks
  Measurement of skin wrinkling depth (px) was evaluated at the crow's feet region and changes were analyzed and digitally photographed in all patients by VisioFace® 1000D (equipped with a high-resolution reflex camera)
R0= Skin firmness (mm) | 6 weeks
  R0 was used as a measure of skin firmness (mm), assessed at the crow's feet region. A Cutometer® dual MPA 580 (Courage & Khazaka) was used to assess skin biomechanical properties
R2= gross elasticity (%) of the skin | 6 weeks
  R2 was used as measure of skin gross elasticity (%), assessed at the crow's feet region. A Cutometer® dual MPA 580 (Courage & Khazaka) was used to assess skin biomechanical properties
R5= Skin net elasticity (%) | 6 weeks
  R5 was used as measure of skin net elasticity (%), assessed at the crow's feet region. A Cutometer® dual MPA 580 (Courage & Khazaka) was used to assess skin biomechanical properties
R7= Skin elastic recovery (%) | 6 weeks
  R7 was used as a measure of skin elastic recovery (%), assessed at the crow's feet region. A Cutometer® dual MPA 580 (Courage & Khazaka) was used to assess skin biomechanical properties
R9= Skin fatigue (mm) | 6 weeks
  R9 was used as a measure of skin fatigue (mm), assessed at the crow's feet region, so a Cutometer® dual MPA 580 (Courage & Khazaka) was used to assess skin biomechanical properties
Skin hydration (AU) | 6 weeks
  Measurement of skin hydration (AU) of the stratum corneum was performed at each study visit by the electrical capacitance method using a Corneometer® CM 825 (Courage & Khazaka, Cologne, Germany).

SECONDARY OUTCOMES:
Subjective perception of product efficacy | At (T6), six weeks after the trial began
  After 6 weeks of treatment, the volunteers filled out questionnaires, to subjectively assess their perception of efficacy. A 3-point Likert scale with the following items: Dissatisfied, slightly satisfied and very satisfied, was used.
Subjective perception of the organoleptic characteristics of the product | At (T6), six weeks after the trial began
  After 6 weeks of treatment, the volunteers filled out questionnaires, to subjectively assess their subjective perception of the organoleptic properties. A 3-point Likert scale with the following items: Dissatisfied, slightly satisfied and very satisfied, was used.
Opinion on the degree of satisfaction with the product | At (T6), six weeks after the trial began
  After 6 weeks of treatment, the volunteers filled out questionnaires, to subjectively evaluate their level of satisfaction with the product. A 3-point Likert scale with the following items: Dissatisfied, slightly satisfied and very satisfied, was used.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Antonio Carrillo, Principal Investigator — University of Extremadura; Rafael Guerrero, Principal Investigator — University of Extremadura
Locations (1):
- GALA Laboratories, Don Benito, Badajoz, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tobin DJ. Introduction to skin aging. J Tissue Viability. 2017 Feb;26(1):37-46. doi: 10.1016/j.jtv.2016.03.002. Epub 2016 Mar 14. PMID 27020864
- [Background] de Miranda RB, Weimer P, Rossi RC. Effects of hydrolyzed collagen supplementation on skin aging: a systematic review and meta-analysis. Int J Dermatol. 2021 Dec;60(12):1449-1461. doi: 10.1111/ijd.15518. Epub 2021 Mar 20. PMID 33742704
- [Background] Wang H. A Review of the Effects of Collagen Treatment in Clinical Studies. Polymers (Basel). 2021 Nov 9;13(22):3868. doi: 10.3390/polym13223868. PMID 34833168
- [Background] Shenoy M, Abdul NS, Qamar Z, Bahri BMA, Al Ghalayini KZK, Kakti A. Collagen Structure, Synthesis, and Its Applications: A Systematic Review. Cureus. 2022 May 9;14(5):e24856. doi: 10.7759/cureus.24856. eCollection 2022 May. PMID 35702467
- [Background] Lupu MA, Gradisteanu Pircalabioru G, Chifiriuc MC, Albulescu R, Tanase C. Beneficial effects of food supplements based on hydrolyzed collagen for skin care (Review). Exp Ther Med. 2020 Jul;20(1):12-17. doi: 10.3892/etm.2019.8342. Epub 2019 Dec 17. PMID 32508986
- [Background] Ryu HS, Joo YH, Kim SO, Park KC, Youn SW. Influence of age and regional differences on skin elasticity as measured by the Cutometer. Skin Res Technol. 2008 Aug;14(3):354-8. doi: 10.1111/j.1600-0846.2008.00302.x. PMID 19159383
- [Background] Pu SY, Huang YL, Pu CM, Kang YN, Hoang KD, Chen KH, Chen C. Effects of Oral Collagen for Skin Anti-Aging: A Systematic Review and Meta-Analysis. Nutrients. 2023 Apr 26;15(9):2080. doi: 10.3390/nu15092080. PMID 37432180
- [Background] Bolke L, Schlippe G, Gerss J, Voss W. A Collagen Supplement Improves Skin Hydration, Elasticity, Roughness, and Density: Results of a Randomized, Placebo-Controlled, Blind Study. Nutrients. 2019 Oct 17;11(10):2494. doi: 10.3390/nu11102494. PMID 31627309
- [Background] Choi FD, Sung CT, Juhasz ML, Mesinkovsk NA. Oral Collagen Supplementation: A Systematic Review of Dermatological Applications. J Drugs Dermatol. 2019 Jan 1;18(1):9-16. PMID 30681787
- [Background] Asserin J, Lati E, Shioya T, Prawitt J. The effect of oral collagen peptide supplementation on skin moisture and the dermal collagen network: evidence from an ex vivo model and randomized, placebo-controlled clinical trials. J Cosmet Dermatol. 2015 Dec;14(4):291-301. doi: 10.1111/jocd.12174. Epub 2015 Sep 12. PMID 26362110
- [Background] Proksch E, Segger D, Degwert J, Schunck M, Zague V, Oesser S. Oral supplementation of specific collagen peptides has beneficial effects on human skin physiology: a double-blind, placebo-controlled study. Skin Pharmacol Physiol. 2014;27(1):47-55. doi: 10.1159/000351376. Epub 2013 Aug 14. PMID 23949208